CLINICAL TRIAL: NCT06936501
Title: Evaluation of the Perception of Freshness and Swallowing Safety in Stroke Patients With Dysphagia Receiving a Specially Designed Thickened Oral Nutritional Supplement: the Cooling Sensation Safe Deglution Study
Brief Title: The Cooling Sensation Safe Deglution Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fundación Pública Andaluza para la Investigación de Málaga en Biomedicina y Salud (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEGLUCOOLING
Record Dates: First submitted 2025-04-14; First posted 2025-04-20 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: Neuromotor Dysphagia After Acute Stroke
Keywords: dysphagia; cerebrovascular accident; oral nutritional supplements
MeSH Terms: conditions — Deglutition Disorders; Stroke

STUDY DESIGN:
Intervention Model Description: Patients will be randomized in a 1:1 ratio
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- GROUP TR (Traditional-->Refreshing) (Active Comparator)
  Interventions: Dietary Supplement: Traditional flavor ONS (vanilla or strawberry, by choice)
- GROUP RT (Refreshing-->Traditional) (Active Comparator)
  Interventions: Dietary Supplement: Refreshing and stimulating flavor ONS (mango-peppermint or lemon-mint, by choice)

INTERVENTIONS:
Dietary Supplement: Traditional flavor ONS (vanilla or strawberry, by choice) — Receives a traditional flavor ONS (vanilla or strawberry, by choice) on days 1 and 2, then switches to a refreshing and stimulating flavor ONS (mango-peppermint or lemon-mint, by choice) on days 3 and 4.
  Arms: GROUP TR (Traditional-->Refreshing)
Dietary Supplement: Refreshing and stimulating flavor ONS (mango-peppermint or lemon-mint, by choice) — Receives a refreshing and stimulating flavor ONS (mango-peppermint or lemon-mint, by choice) on days 1 and 2, then switches to a traditional flavor ONS (vanilla or strawberry, by choice) on days 3 and 4.
  Arms: GROUP RT (Refreshing-->Traditional)

SUMMARY:
Dysphagia is a common complication in patients who have suffered a cerebrovascular accident (CVA), with an incidence ranging from 29% to 81%. Rehabilitation improves dysphagia in 47% of cases within the first few weeks and in 17% within 2-4 months. However, dysphagia can lead to nutritional and respiratory complications, affecting recovery and increasing healthcare costs due to the need for prolonged hospitalizations and readmissions.

Malnutrition is a frequent consequence of CVA, with its prevalence increasing from 12% to 50% in patients with prolonged hospital stays. This condition worsens the vital prognosis, as it increases the incidence of complications and slows down functional recovery.

Post-stroke dysphagia causes unsafe swallowing and increases the risk of aspiration, pneumonia, and other respiratory infections, worsening the patient's prognosis. Impaired swallowing efficiency leads to oral and pharyngeal residue, aggravating nutritional complications. On the other hand, swallowing safety is characterized by the presence of aspirations, manifesting as coughing, wet voice, and oxygen desaturation during the Volume-Viscosity Swallow Test (V-VST).

The dietary management of these patients includes modifying food textures and using thickened liquids, strategies that have been shown to reduce the incidence of aspiration pneumonia. However, adherence to these diets is often low due to dissatisfaction with the texture and taste of thickening agents.

In this context, the development of oral nutritional supplements (ONS) with stimulating flavors has been proposed to improve the perception of swallowing safety. Stimulation of the oropharyngeal sensory nerves, through activation by cold and chemical agents such as menthol, enhances swallowing by increasing oral sensitivity and improving the pharyngeal swallowing reflex response. The European Society for Swallowing Disorders (ESSD) recommends sensory stimulation as a therapeutic strategy to compensate for oropharyngeal sensory loss in patients with dysphagia.

Previous studies have shown that sensory stimulation activates the swallowing center in the brainstem, accelerating the swallowing response and protecting the airway. In clinical trials with transient receptor potential (TRP) receptor agonists, observed benefits include faster closure of swallowing sphincters, improved swallowing reflex sensitivity, a 50% reduction in microaspirations, and a 67% decrease in pharyngeal residue.

Based on this evidence, a new thickened ONS with stimulating flavors such as mango-mint and lemon-mint has been designed to enhance the perception of freshness and swallowing safety. This supplement is already used in clinical practice, but its effect on the perception of patients with post-stroke dysphagia has not yet been evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Men and women over 18 years old.
* Currently hospitalized due to an acute stroke.
* Confirmed diagnosis of dysphagia through V-VST (Volume-Viscosity Swallow Test).
* Ability to collaborate and respond to questionnaire questions and other research tools used in the study.
* Malnutrition or risk of malnutrition, requiring a thickened, high-calorie, high-protein ONS, as determined by medical assessment in routine clinical practice.
* Voluntary written informed consent to participate in the study.

Exclusion Criteria:

* Moderate to severe cognitive impairment that interferes with the correct interpretation of the study or its requirements.
* Diagnosis of advanced dementia, severe psychiatric illness, or any other central nervous system condition that impairs the patient's comprehension of the study.
* Sociocultural, linguistic, intellectual, or other factors that hinder the patient's proper understanding of the study.
* Diagnosis of galactosemia.
* Intolerance or refusal (for any reason) of oral nutritional supplements.
* Requirement for parenteral nutrition or contraindication to oral intake.
* Severe active renal, hepatic, or gastrointestinal diseases that contraindicate the use of ONS

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Perception of swallowing safety of thickened ONS | At 48 and 96 hours
  Objective: To assess the perceived safety when swallowing based on the flavor of the thickened ONS.
  * Ad hoc questionnaire , designed exclusively for this study
  * Two closed-ended questions
  * Response scale: Visual Numeric Scale (VNS) from 0 to 10
  * 0 = No sensation of safety
  * 10 = Maximum sensation of safety
  * Based on previously used scales in healthy individuals
Assessment using selected items from the validated Spanish version of the EAT-10 scale | At 48 and 96 hours
  * Items focused on perceived safety during swallowing:
  * Item 8: "When I swallow, food sticks in my throat."
  * Item 9: "I cough when I eat."
  * Item 10: "Swallowing is stressful." Responses are scored from 0 to 4, where 0 = no problem; 4 = severe problem This scale is validated in Spanish. The combination of a validated scale and an ad hoc scale seeks to strengthen the study's methodological robustness.
Perception of freshness of thickened ONS | At 48 and 96 hours
  Objective: To assess the perception of freshness that stimulates swallowing, depending on the flavor of the thickened ONS received.
  * Ad hoc questionnaire , designed exclusively for this study
  * Three closed-ended questions
  * Response scale: Visual Numeric Scale (VNS) from 0 to 10
  * 0 = No freshness
  * 10 = Maximum sensation of freshness
  * Based on scales used previously in healthy subjects

SECONDARY OUTCOMES:
Evaluation of Satisfaction of thickened ONS | At 48 and 96 hours
  Objective: To assess patient satisfaction with the thickened ONS.
  * Ad hoc questionnaire , designed exclusively for this study
  * Based on statements related to:
  * Safety
  * Texture
  * Mouthfeel
  * Overall satisfaction
  * 5-point Likert scale:
  * 1 = Not at all
  * 5 = Very much
Evaluation of Tolerability of thickened ONS | At 48 and 96 hours
  Objective: To assess perceived tolerability of the thickened ONS.
  * Ad hoc questionnaire, designed exclusively for this study
  * Includes 7 closed-ended questions
  * Visual Numeric Scale (VNS) from 0 to 10:
  * 0 = Not tolerable at all
  * 10 = Fully tolerable
Evaluation of Consumption of thickened ONS | At 48 and 96 hours
  Objective: To record the amount of thickened ONS consumed compared to the medical recommendation.
  * Ad hoc questionnaire (not validated), designed exclusively for this study
  * Patient's intake percentage:
  * 100%, 75%, 50%, 25%, 0%
  * If <50% was consumed, patients will indicate one or more of the following reasons:
  * TASTE is unpleasant
  * SMELL is unpleasant
  * TEXTURE is unpleasant
  * APPEARANCE is unpleasant
  * VOLUME is too much
  * Poor TOLERANCE
  * FEAR of swallowing
  * PAIN when swallowing
  * FORGOT to take it

CONTACTS AND LOCATIONS:
Overall Officials: Gabriel Olveira Fuster, PhD, MD, Principal Investigator — Hospital Regional de Malaga
Locations (1):
- Hospital Regional Universitario de Málaga, Málaga, Málaga, Spain